CLINICAL TRIAL: NCT00653107
Title: Palliation of Dysphagia in Patients With Advanced Cancer of the Oesophagus by Comparing Stent Followed by 3 Courses of Brachytherapy With 3 Courses of Brachytherapy Only. A Randomised Phase III Study (PACO)
Brief Title: Palliation Dysphagia Cancer Oesophagus Stent+Brachytherapy Versus Brachytherapy Only
Acronym: PACO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was closed prematurely due to slow recruitment
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Cecilie Delphin Amdal, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FO2007/45; S-07447a
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Esophageal Neoplasm
Keywords: Palliation; Cancer oesophagus; Stent; Brachytherapy; Randomized
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Stent followed by 3 brachytherapy fractions
  Interventions: Procedure: Stent insertion; Radiation: Brachytherapy
- B (Active Comparator): 3 fractions of brachytherapy
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Procedure: Stent insertion — Self-expanding metal stents will be used. These will be of the type which the hospital at any given time uses, at present Ultraflex®.
  Arms: A
Radiation: Brachytherapy — a flexible applicator (with a diameter adapted to the stent's diameter) will be introduced into the oesophagus, so the applicator will be lying in the middle of the lumen of the stent. Thereafter, the flexible applicator is connected to a MicroSelectron afterloading device (Iridium-192), and the treatment is given with a high dose rate (> 12 Gy/h).
  Arms: A
Radiation: Brachytherapy — a flexible applicator will be introduced into the oesophagus. The flexible applicator is connected to a MicroSelectron afterloading device (Iridium-192), and the treatment is given with a high dose rate (> 12 Gy/h).
  Arms: B

SUMMARY:
We wish to improve the swallowing function of patients with advanced cancer of the oesophagus, by carrying out a randomised clinical study in which we compare primary stenting followed by brachytherapy in the stent, 8 G x 3 with standard brachytherapy 8 Gy x 3.

The aim of the study is to investigate whether patients who receive a stent followed by brachytherapy have a better swallowing function without more pain at week +2,compared to patients who receive brachytherapy alone.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all the following criteria:

1. Histologically or cytologically verified carcinoma of the oesophagus
2. Reduced ability to swallow solid food, minimum grade 1 (see page 16)
3. Age ≥ 18 years
4. Ability to understand and answer (with or without help) the study questionnaires
5. Written informed consent received
6. A Completed questionnaire received from the patient
7. One of the following criteria must be fulfilled:

   1. Advanced disease and WHO performance status ≥2
   2. Advanced disease and WHO performance status 0-1 and other therapy excluded due to medical condition
   3. Advanced disease and WHO performance status 0-1 and patient's preference
   4. Local disease and WHO performance status ≥2 and other therapy excluded due to medical condition
   5. Local disease and WHO performance status ≥2 and patient's preference

Exclusion Criteria:

1. Oesophageal stent already inserted
2. Endoscopic procedures not tolerated
3. Cannot have (additional) radiation therapy
4. Tumour location not suited for stent or brachytherapy (the upper 3 cm of oesophagus or major component in the cardia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dysphagia measured with the dysphagia grading scale at week +2 after start of treatment. Pain at rest measured with ESAS at week +2 after start of treatment. | 8 years

SECONDARY OUTCOMES:
Health related quality of life | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bjordal, PhD, Principal Investigator — Radiumhospitalet. Rikshospitalet HF
Locations (1):
- Radiumhospitalet, Oslo, Norway